CLINICAL TRIAL: NCT06522984
Title: Fractional Erbium YAG Laser vs Intradermal and Systemic Tranexamic Acid in Combination With Topical Hydroquinone for Refractory Melasma
Brief Title: Fractional Erbium YAG Laser vs Intradermal and Systemic Tranexamic Acid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Aswan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Heba Allah Mohamed Mustafa
Record Dates: First submitted 2024-07-15; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-06

CONDITIONS: Refractory Melasma
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): About 15 cases will receive sessions with fractional Er: YAG laser every 3 weeks followed by application of topical 4% (HQ) cream.
  Interventions: Drug: Tranexamic acid injection
- Group B (Active Comparator): About 15 cases will receive sessions of intradermal injection of tranexamic acid on the melasma site every 3 weeks concurrently with the application of topical 4% HQ cream every night. The injections will be done using an insulin syringe with a dilution of the tranexamic acid
  Interventions: Drug: Tranexamic acid injection
- Group C (Active Comparator): About 15 cases will receive oral tranexamic acid 500mg tablet once daily for three months. And will also be asked to apply a thin layer of topical HQ 4% cream on the hyperpigmented areas once every night.
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — to evaluate and compare efficacy of:
  * Fractional Er: YAG laser combined with topical hydroquinone.
  * Intradermal injection of tranexamic acid combined with topical hydroquinone cream.
  * Oral administration of tranexamic acid combined with topical hydroquinone cream. In treating refractory melasma.
  Other Names: Fractional erbium YAG laser

SUMMARY:
Melasma is a common acquired disorder of hyperpigmentaion caused by increased melanin production by melanocytes.

Melasma is a name derived from the Greek word melas meaning black.It is characterized by the appearance of brownish or grayish symmetrical patches on sun-exposed skin, most commonly on the face. Compared to men, women are more likely to be affected.

DETAILED DESCRIPTION:
Melasma is more common in people with dark complexions and Fitzpatrick skin types III IV.Depending on ethnicity and region, melasma prevalence might vary from 8.8% to 40%. The cause of melasma is still unknown in the meantime.

Numerous elements, including genetics, sunshine, endocrine stimulation, oxidative conditions,pregnancy, exogenous hormons,and morphofunctional changes, may have a role in the development of the disease.

Since melasma is a common skin condition affecting mostly pregnant women and those on hormonal birth control, it is known as the "mask of pregnancy,

Treatment for melasma remains a challenge, with substantial psychosocial ramifications. Many factors, including variability in clinical presentation and responsiveness to treatment between genders, skin phototypes, and ethnicities, can affect treatment efficacy. None of variety methods have been sufficiently effective to be considered the gold standard.

Hydroquinone (HQ) has historically been the most studied topical agent in the treatment of melasma. HQ is a hydroxyphenolic compound that inhibits the conversion of dopa to melanin by the inhibition of tyrosinase; it also inhibits RNA and DNA synthesis of melanocytes and degrades melanosomes.

Tranexamic acid (TXA) is an antifibrinolytic drug that has been used off-label for the treatment of melasma, as an oral or intradermal injection.

TXA is a lysine-derived amino acid with anti-inflammatory effects that prevents ultraviolet (UV)-induced skin pigmentation by inhibiting attachment of plasminogen to keratinocytes and activation of plasmin. Plasmin stimulates melanogenesis by conversionof arachidonic acid to prostaglandin and leukotriene. On the other hand, plasmin increases the level of melanogenic factors.

Laser therapy is a unique ablative modality that might potentially increase the penetration of medications applied topically by destroying the SC, epidermal, and dermal layers of the skin in a predictable and controlled manner.

The Fractional erbiumdoped yttrium aluminum garnet (Er: YAG) laser has a wavelength of 2,940 nm and is strongly absorbed by water in the epidermis. It exerts its ablation effect with minimal penetration depth and minimal heat generation and therefore minimal thermal damage.

ELIGIBILITY:
Inclusion Criteria:

- Patients of both sexes with melasma.

Exclusion Criteria:

* Pregnancy
* Lactation
* Administration of oral contraceptive pills or any phototoxic drug within 1 month prior to study
* Patients with a history of thrombosis, abnormal bleeding profile, known hypersensitivity to TA or HQ, and endocrinal disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Refractory Melasma Treatment combination with topical hydroquinone | 3 months
  to detect the treatment response by YAG laser vs intradermal and systemic tranexamic acid by using The MASI index ( MASI is an index designed to quantify the severity of melasma during therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Adam Ali El Taieb, Professor, Study Chair — Dermatology, Venereology and Andrology.Faculty of Medicine, Aswan University
Locations (1):
- Aswan University hospitals, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided